CLINICAL TRIAL: NCT03096938
Title: Cell-free DNA Methylation Markers for Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Prof., Sun Yat-sen University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: cancer screening
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Cancer Screening
Keywords: cell-free DNA; methylation; markers; cancer; screening
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal screening group (Placebo Comparator): patients receive the routine screening examination
  Interventions: Diagnostic Test: methylation markers screening
- methylation markers screening group (Experimental): patients receive the methylation markers screening
  Interventions: Diagnostic Test: methylation markers screening

INTERVENTIONS:
Diagnostic Test: methylation markers screening — Cell-free DNA extraction from plasma samples-Bisulfite conversion of cfDNA-Determination of DNA methylation levels by deep sequencing-Sequencing data analysis

SUMMARY:
The purpose of this study is to evaluate the role of cell-free DNA methylation markers in cancer screening.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is average risk for development of cancer
2. Subject able and willing to undergo screening test within 90 days of enrollment
3. Subject is 40 to 74 years of age inclusive
4. Subject is able to comprehend, sign, and date the written informed consent document to participate in the study

Exclusion Criteria:

1. Subject has any condition which, in the opinion of the investigator should preclude participation in the study
2. Subject has a history of cancer
3. Participation in any "interventional" clinical study within the previous 30 days in which an experimental treatment is administered or might be administered through a randomized assignment of the subject to one or more study groups.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity (true positive rate) | 2 year
  The proportion of persons with disease who have a positive test (positive test results among persons with disease)
Specificity (true negative rate) | 2 year
  The proportion of persons without disease who have a negative test (negative test results among persons without disease)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Imperiale TF, Ransohoff DF, Itzkowitz SH, Levin TR, Lavin P, Lidgard GP, Ahlquist DA, Berger BM. Multitarget stool DNA testing for colorectal-cancer screening. N Engl J Med. 2014 Apr 3;370(14):1287-97. doi: 10.1056/NEJMoa1311194. Epub 2014 Mar 19. PMID 24645800